CLINICAL TRIAL: NCT04345952
Title: Can a Mindfulness Meditation App Reduce Emotional Distress in Colorectal Cancer Patients Undergoing Adjuvant Chemotherapy
Brief Title: Calm for Cancer Patients Receiving Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never submitted to the IRB so never received permission to or enrolled any subjects
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTMS# 20-0117; HSC20200636H (Other: UT Health Science Center San Antonio IRB)
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-12

CONDITIONS: Cancer Colorectal
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calm Meditation (Experimental): Participants in the Calm group will be asked to use the Calm app ad libitum during their time spent receiving chemotherapy at the Mays Cancer Center (~2 hours) and while at home between treatment cycles ad libitum. Participation will be measured during the entire intervention using internal tracking systems within the app (i.e., # of times logged in, type of meditation accessed, time spent meditating, date and time of meditation accessed). This data will be provided to us through data coordinator of the app.
  Interventions: Behavioral: Calm Meditation Mobile App
- Usual Care (No Intervention): The usual care control group will not be offered anything to listen to during their chemotherapy treatment cycles or when they are between chemotherapy treatment cycles. They will receive their treatment as intended without any additional intervention.

INTERVENTIONS:
Behavioral: Calm Meditation Mobile App — The Calm Meditation Mobile App will be used to deliver the meditation intervention to study participants. The Calm app is downloaded onto the participant's smartphone.
  Arms: Calm Meditation

SUMMARY:
Chemotherapy is a common strategy used to treat colorectal cancer patients, but is often leads patients and survivors to experience a host of symptoms, of which acute emotional distress is a major concern. Smartphone-based meditation via an already-developed app (i.e., Calm) is a unique and novel way of providing a potentially helpful symptom-management strategy to colorectal cancer patients and survivors both during their chemotherapy treatment sessions for the management of distress and between treatment sessions for the management of other more chronic symptoms. Our hypothesis is that colorectal cancer patients using the Calm smartphone app throughout their chemotherapy treatment will see lower psychological distress during individual chemotherapy treatment sessions, greater chemotherapy tolerability, lower chemotherapy toxicity symptoms, lesser fatigue, and higher quality of life as compared to a usual care control group. Colorectal cancer patients (N=30) will be randomly assigned to an intervention (n=15) or control group (n=15) for the duration of their chemotherapy treatment, with study outcome measurement occurring throughout their treatment.

DETAILED DESCRIPTION:
Chemotherapy is a common treatment modality among colorectal cancer patients. Despite improvements in survival among those receiving chemotherapy, patients often experience side effects including pain, nausea, vomiting, changes in appetite and weight, fatigue, depressed mood, and reduced quality of life. Colorectal cancer patients undergoing chemotherapy also experience acute elevation in psychological distress (e.g., anxiety, stress). Worldwide, as many as 40% of cancer patients currently report using complementary and alternative medicine (CAM) for the management of their diagnosis and treatment-related side effects. Evidence to support the efficacy of various CAM approaches is still in its infancy, and further research is warranted.

Mindfulness-based strategies, a popular CAM approach among cancer patients, may have unique benefits for addressing both treatment-related side effects as well as the management of acute levels of psychological distress experienced while undergoing chemotherapy. Preliminary evidence supports the benefits of meditation, relaxing sounds, and progressive muscle relaxation for the reduction of distress and state anxiety as well as the improvement of neuroendocrine responses, indicative of improved stress response, among cancer patients undergoing chemotherapy. Additionally, meditation has been shown to improve distress, cognitive function, mental health, quality of life, and chemotherapy-related neurotoxicity symptoms among cancer patients that had undergone chemotherapy treatment. Despite preliminary evidence to support mindfulness-based strategies to help cancer patients undergoing chemotherapy, further research is needed to determine their efficacy.

Smartphone applications (apps) are a unique mode of delivering mindfulness-based strategies to cancer patients and may help make CAM more accessible to cancer patients reporting barriers to participation in in-person interventions (e.g., pain, fatigue, transportation, scheduling difficulties, etc.). Additionally, smartphone apps are a way of providing mindfulness-based strategies to patients while undergoing chemotherapy without the need of specialized personnel to lead mindfulness-based sessions for patients in the clinic. Smartphone accessibility is becoming more ubiquitous, with nearly three quarters of cancer patients reporting access to a mobile smartphone. To our knowledge there have been no studies that have tested the effects of meditation delivered specifically via a smartphone app to cancer patients undergoing chemotherapy (one study used an iPad). The investigators have previously demonstrated the feasibility and preliminary effects of delivering four weeks of smartphone-based meditation (via the Calm app) to hematological cancer patients to improve symptom burden. However, these patients were not undergoing chemotherapy. A meditation app such as Calm could be used to deliver mindfulness-based strategies to cancer patients undergoing chemotherapy while in clinic and outside of clinic for the management of acute psychological distress and chemotherapy-related side effects.

The Calm app has over 2 million paying users and 65 million downloads, and was named Apple's "App of the Year" in 2017.9,10 The Calm app was developed based on tenets of mindfulness and cognitive behavioral therapy, and provides its users with a range of mindfulness-based options to choose from, including meditations, Sleep Stories, and Soundscapes. In the proposed study, the investigators will investigate the use of Calm among a small sample of colorectal cancer patients (N=30; n=15 per group) who are beginning adjuvant chemotherapy within 12-weeks post-surgery as compared to a usual care control group to determine its effects on acute psychological distress within a single chemotherapy session as well as chemotherapy-related side effects.

STUDY OBJECTIVES

Objective 1: Investigate the effects of using a meditation app to reduce psychological distress (measured using the Distress Thermometer), across multiple chemotherapy sessions (n=15) among colorectal cancer patients as compared to usual control (n=15).

The primary hypothesis for this objective is that those using a meditation app will experience a reduction in psychological distress from beginning to end of each chemotherapy session as compared to usual care.

Objective 2: Investigate the effects of using a meditation app on chemotherapy toxicity and tolerability (measured using patient medical records; dose reduction/modification, dose delays, # of cycles completed, hospitalization, cytopenias, etc.), fatigue (measured using the Brief Fatigue Inventory), and quality of life (measured using the General Version of the Functional Assessment of Cancer and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) among colorectal cancer patients during a chemotherapy treatment cycle (i.e., two-three week cycle between the sessions) as compared to a usual care control group.

The primary hypothesis for this objective is that those using the meditation app will experience less severe chemotherapy toxicity, greater chemotherapy tolerability, less fatigue, and greater quality of life as compared to the usual care control group.

ELIGIBILITY:
Inclusion Criteria:

* Have a colorectal cancer diagnosis and waiting the beginning of adjuvant chemotherapy treatment at the Mays Cancer Center University of Texas (UT) Health San Antonio
* Own a mobile smartphone (iPhone with iOS 9.0 or later or an Android 4.1 or later)
* Willing to download a mobile app
* Able to read and understand English or Spanish
* Aged 18 years or older
* Willing to be randomized to one of two groups

Exclusion Criteria:

* Meditation or meditative movement practice (i.e., yoga, tai chi, qigong) of greater than or equal to 60 min/month in the past six months
* Use of any consumer-based meditation app
* Reside outside of the united states

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Distress | 6-month average change from baseline (beginning of chemotherapy treatment session) to post-treatment (end of chemotherapy treatment session)
  Distress will be measured with the Distress Thermometer at the beginning and end of each chemotherapy treatment session over the course of the approximate 6-month study duration. The Distress Thermometer is a 10-point visual analog scale and a higher score indicates greater distress.

SECONDARY OUTCOMES:
Chemotherapy toxicity and tolerability | Post-intervention (month 6)
  Chemotherapy toxicity and tolerability will be assessed through patient medical records by pulling the following variables from their record: dose reduction/modification, dose delays, # of cycles completed, hospitalization, cytopenias
Change in Fatigue | Change from baseline (week 0) to post-intervention (month 6)
  Fatigue will be measured with the Brief Fatigue Inventory (BFI). The score on the BFI ranges from 0-90 with a higher score indicating a higher amount of fatigue being measured.
Change in Cancer Treatment-Related Quality of Life | Change from baseline (week 0) to post-intervention (month 6)
  Cancer Treatment-Related Quality of Life will be measured with the General Version of the Functional Assessment of Cancer. The Scale is scored on a 0-100 normalized scale with a higher score indicating a higher quality of life.
Change in Cancer Health-Related Quality of Life | Change from baseline (week 0) to post-intervention (month 6)
  Cancer Health-Related Quality of Life will be measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. The scale scoring ranges from 0-100 with a higher score indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Mesa, Principal Investigator — Mays Cancer Center at UT Health San Antonio MD Anderson
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No